CLINICAL TRIAL: NCT02091999
Title: A Phase 1 Study of the Safety and Pharmacokinetics of Escalating Doses of ASG-22CE Given as Monotherapy in Subjects With Metastatic Urothelial Cancer and Other Malignant Solid Tumors That Express Nectin-4
Brief Title: A Study of Escalating Doses of ASG-22CE Given as Monotherapy in Subjects With Metastatic Urothelial Cancer and Other Malignant Solid Tumors That Express Nectin-4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASG-22CE-13-2
Expanded Access: NCT04136808 (Approved for marketing)
Record Dates: First submitted 2014-03-18; First posted 2014-03-19 (Estimated); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Urothelial Cancer and Other Malignant Solid Tumors
Keywords: enfortumab vedotin; Metastatic Urothelial Cancer; Safety; AGS-22C3E; EV-101; Nectin 4 protein, humans; Clinical Trial, Phase 1; ASG-22CE; ASG-22ME; Pharmacokinetics of ASG-22CE
MeSH Terms: interventions — enfortumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A enfortumab vedotin Dose Escalation (Dose Levels 1-4) (Experimental): All subjects will receive a single 30 minute intravenous (IV) infusion of enfortumab vedotin once weekly for the first 3 weeks of every 4 week cycle (i.e., on Days 1, 8 and 15).
  Interventions: Drug: enfortumab vedotin
- Part B enfortumab vedotin Renal Insufficiency Expansion (Experimental): Subjects will receive a single 30 minute IV infusion of enfortumab vedotin at a dose level below and escalated up to the preliminary RP2D once weekly for 3 weeks of every 4 weeks (i.e., on Days 1, 8 and 15) until disease progression, intolerability of the investigational product or consent withdrawal. A cycle is 4 weeks.
  Interventions: Drug: enfortumab vedotin
- Part B enfortumab vedotin NSCLC Expansion (Experimental): Subjects will receive a single 30 minute IV infusion of enfortumab vedotin at the preliminary RP2D once weekly for 3 weeks of every 4 weeks (i.e., on Days 1, 8 and 15) until disease progression, intolerability of the investigational product or consent withdrawal. A cycle is 4 weeks.
  Interventions: Drug: enfortumab vedotin
- Part B enfortumab vedotin Ovarian Cancer Expansion (Experimental): Subjects will receive a single 30 minute IV infusion of enfortumab vedotin at the preliminary RP2D once weekly for 3 weeks of every 4 weeks (i.e., on Days 1, 8 and 15) until disease progression, intolerability of the investigational product or consent withdrawal. A cycle is 4 weeks.
  Interventions: Drug: enfortumab vedotin
- Part C enfortumab vedotin CPI Treated Expansion (Experimental): Subjects will receive a single 30 minute IV infusion of enfortumab vedotin at the preliminary RP2D once weekly for 3 weeks of every 4 weeks (i.e., on Days 1, 8 and 15). A cycle is 4 weeks. Subjects will continue treatment until disease progression, intolerability of enfortumab vedotin, Investigator decision or consent withdrawal.
  Interventions: Drug: enfortumab vedotin

INTERVENTIONS:
Drug: enfortumab vedotin — intravenous (IV) infusion
  Other Names: ASP7465; ASG-22CE; ASG-22ME

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics of enfortumab vedotin as well as assess the immunogenicity and antitumor activity in subjects with metastatic urothelial cancer and other malignant solid tumors that express Nectin-4.

DETAILED DESCRIPTION:
All subjects will receive a single 30 minute IV infusion of enfortumab vedotin once weekly for the first 3 weeks of every 4 weeks (i.e., on Days 1, 8, and 15). A cycle is 4 weeks.

This is a 3 part study. Part A will evaluate enfortumab vedotin in subjects with histologically confirmed malignant solid tumors (excluding sarcomas) that are resistant or have recurred. Subjects will continue treatment until disease progression, intolerability of enfortumab vedotin, investigator decision or consent withdrawal. Part A will follow a modified Continual Reassessment Method (mCRM).

Part B, will evaluate enfortumab vedotin in 3 different expansion cohorts: 1) Urothelial cancer subjects with renal insufficiency defined as a Creatinine Clearance ≥ 15 ml/min and < 30 ml/min, 2) subjects with Metastatic Non Small Cell Lung Cancer (NSCLC) and 3) subjects with Metastatic Ovarian Cancer. With the exception of the renal insufficiency cohort, enrollment into Part B will occur at the recommended phase 2 dose (RP2D) established in Part A. Enrollment into the renal insufficiency cohort will begin at starting dose and escalated using a 3 + 3 dose escalation design. Subjects will continue treatment until disease progression, intolerability of enfortumab vedotin or consent withdrawal.

Part C will evaluate enfortumab vedotin at the RP2D (determined from Part A) in subjects who have been previously treated with immune checkpoint inhibitors (CPI) in the metastatic setting. Subjects will continue treatment until disease progression, intolerability of enfortumab vedotin, investigator decision or consent withdrawal.

All subjects will be followed post-treatment through the 30-day Safety Follow-up Visit.

ELIGIBILITY:
Inclusion Criteria:

* Dose Escalation, Renal insufficiency and CPI-Treated Expansion cohorts: Histologically confirmed Transitional Cell Carcinoma of the Urothelium (TCCU) (i.e., cancer of the bladder, renal pelvis, ureter, or urethra). Subjects with Urothelial Carcinoma with squamous differentiation or mixed cell types are eligible.
* Ovarian Expansion Cohort: Subjects with recurrent disease or histologically or cytologically confirmed Stage III/IV diagnosis of epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal carcinoma who have previously progressed while receiving or within 6 months of completing a platinum-containing regimen.
* NSCLC Expansion Cohort: Histologic or cytologic diagnosis of NSCLC (squamous or non-squamous or NSCLC-not specified)
* Dose Escalation, Renal insufficiency, NSCLC and CPI-Treated Expansion Cohorts: For subjects with urothelial cancer and NSCLC: Subjects must submit a tumor tissue for Nectin-4 expression. Enrollment for these subjects is not dependent on the immunohistochemistry using the H-Score (IHC H-Score).
* Ovarian Expansion Cohort: Subjects must have tumor tissue positive (IHC H-score ≥150) for Nectin-4 expression
* For Dose Escalation, NSCLC and Ovarian Expansion Cohorts: Subject must have failed at least one prior chemotherapy regimen for metastatic disease (urothelial and bladder cancer subjects are not required to have failed prior chemotherapy regimen if considered unfit for cisplatin-based chemotherapy)
* For the CPI-Treated Expansion Cohort: Subject must have received prior treatment with a CPI in the metastatic setting.
* Subjects must have measurable disease according to RECIST (version 1.1)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of ≥ 3 months
* Negative pregnancy test (women of childbearing potential)
* Hematologic function, as follows (no red blood cell or platelet transfusions are allowed within 14 days of the first dose of enfortumab vedotin):

  * Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L
  * Platelet count ≥ 100 x 10^9/L
  * Hemoglobin ≥ 9 g/dL
* Renal function, as follows: Dose Escalation, NSCLC, Ovarian, and CPI Treated Expansion Cohorts: creatinine clearance of ≥ 30 mL/min by the Cockcroft-Gault equation or as measured by 24 hour urine collection. For the Renal Insufficiency Expansion Cohort: creatinine clearance estimate ≥15 ml/min and <30 ml/min by Cockcroft-Gault equation or as measured by 24 hour urine collection.
* Total bilirubin ≤ 1.5 x ULN (upper limit of normal)
* Serum albumin ≥2.5 g/dL
* Aspartate aminotransferase (AST) ≤ 1.5 x ULN
* Alanine aminotransferase (ALT) ≤ 1.5 x ULN
* International normal ratio (INR) < 1.3 or ≤ institutional ULN (or ≤ 3.0 if on therapeutic anticoagulation)
* Sexually active fertile subjects, and their partners, must agree to use medically accepted double-barrier methods of contraception (e.g., barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the study and at least 6 months after termination of study therapy
* Competent to comprehend, sign, and date an independent ethics committee/institutional review board/research ethics board (IEC/IRB/REB) approved informed consent form

Exclusion Criteria:

* Preexisting sensory neuropathy Grade ≥ 2
* Preexisting motor neuropathy Grade ≥ 2
* Uncontrolled central nervous system metastases
* Use of any investigational drug within 14 days prior to the first dose of study drug
* Any anticancer therapy within 14 days prior to the first dose of study drug, including: small molecules, immunotherapy, chemotherapy, monoclonal antibody therapy, radiotherapy or any other agents to treat cancer (anti-hormonal therapy given as adjuvant therapy for early-stage estrogen receptor (ER) positive breast cancer is not considered cancer therapy for the purpose of this protocol)
* Subjects with immunotherapy related adverse events requiring high doses of steroids (≥ 40 mg/day of prednisone) are not eligible.
* Any P-glycoprotein (P-gp) inducers/inhibitors or strong cytochrome P4503A (CYP3A) inhibitors within 14 days prior to the first dose of study drug
* Thromboembolic events and/or bleeding disorders ≤ 14 days (e.g., deep vein thrombosis (DVT) or pulmonary embolism (PE)) prior to the first dose of study drug
* Documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms (including congestive heart failure) consistent with New York Heart Association Class III-IV within 6 months prior to the first dose of enfortumab vedotin.
* Known Human Immunodeficiency Virus (HIV) or Acquired Immune Deficiency Syndrome (AIDS)
* Subjects with a positive Hepatitis B surface antigen and/or antihepatitis B core antibody. Subjects with a negative polymerase chain reaction (PCR) assay are permitted with appropriate antiviral prophylaxis.
* Active Hepatitis C infection. Subjects who have been treated for Hepatitis C infection can be included if they have documented sustained virologic response of ≥ 12 weeks.
* Decompensated liver disease as evidenced by clinically significant ascites refractory to diuretic therapy, hepatic encephalopathy, or coagulopathy
* Known sensitivity to any of the ingredients of the investigational product enfortumab vedotin (ASG-22CE)
* Major surgery within 28 days prior to first dose of study drug
* History of another malignancy within 3 years before the first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy. Subjects with nonmelanoma skin cancer, localized prostate cancer treated with curative intent with no evidence of progression, low-risk or very low risk localized prostate cancer under active surveillance/watchful waiting without intent to treat, or carcinoma in situ of any time (if complete resection was performed) are allowed.
* History of uncontrolled diabetes mellitus or diabetic neuropathy within 3 months of the first dose of study drug. Uncontrolled diabetes is defined as hemoglobin A1C (HbA1c) ≥ 8% or HbA1c > 7 to < 8% with associated diabetes symptoms (polyuria or polydipsia) that are not otherwise explained.
* Currently receiving systemic antimicrobial treatment for active infection (viral, bacterial, or fungal) at the time of first dose of enfortumab vedotin. Routine antimicrobial prophylaxis is permitted.
* Condition or situation which may put the subject at significant risk, may confound the study results, or may interfere significantly with subject's participation in the study
* Any medical, psychiatric, addictive or other kind of disorder which compromises the ability of the subject to give written informed consent and/or to comply with procedures
* Has ocular conditions such as:

  * Active infection or corneal ulcer (e.g. keratitis)
  * Monocularity
  * History of corneal transplantation
  * Contact lens dependent (if using contact lens, must be able to switch to glasses during the entire study duration)
  * Uncontrolled glaucoma (topical medications allowed)
  * Uncontrolled or evolving retinopathy, wet macular degeneration, uveitis, papilledema, or optic disc disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2014-05-14 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | up to 36 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE): Concentration at the end of infusion (CEOI) | Days 1-4, 8, 15-18 of Cycle 1 and Days 1, 8, and 15 of Cycle 2 and Day 1 of subsequent cycles up to an average of 24 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE): Maximum observed concentration (Cmax) | Days 1-4, 8, 15-18 of Cycle 1 and Days 1, 8, and 15 of Cycle 2 and Day 1 of subsequent cycles up to an average of 24 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE): Trough concentration (Ctrough) | Days 1-4, 8, 15-18 of Cycle 1 and Days 1, 8, and 15 of Cycle 2 and Day 1 of subsequent cycles up to an average of 24 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE): Time to maximum concentration (Tmax) | Days 1-4, 8, 15-18 of Cycle 1 and Days 1, 8, and 15 of Cycle 2 and Day 1 of subsequent cycles up to an average of 24 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE): Partial area under the serum concentration-time curve after first dose and as appropriate (AUC0-7) | Days 1-4, 8, 15-18 of Cycle 1 and Days 1, 8, and 15 of Cycle 2 and Day 1 of subsequent cycles up to an average of 24 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE): Terminal or apparent terminal half-life (t1/2) | Days 1-4, 8, 15-18 of Cycle 1 and Days 1, 8, and 15 of Cycle 2 and Day 1 of subsequent cycles up to an average of 24 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE): Systemic clearance (CL) | Days 1-4, 8, 15-18 of Cycle 1 and Days 1, 8, and 15 of Cycle 2 and Day 1 of subsequent cycles up to an average of 24 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE): Volume of distribution at steady state (Vss) | Days 1-4, 8, 15-18 of Cycle 1 and Days 1, 8, and 15 of Cycle 2 and Day 1 of subsequent cycles up to an average of 24 months

SECONDARY OUTCOMES:
Incidence of Anti-Drug Antibody (ADA) | up to 24 months
Tumor response | up to 24 months
  Incidence of tumor response defined as either a complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) criteria (version 1.1) that is confirmed ≥ 28 days later
Objective response rate | up to 24 months
  Defined as the percentage of subjects who experience a best response of either CR or PR in that cohort. CR and PR must be confirmed ≥ 28 days later.
Disease control rate | up to 24 months
  Defined as the percentage of subjects who experience a best response of CR, PR or stable disease (SD)
Progression Free Survival (PFS) | 36 months
  Time from the date of first infusion to the earliest date of documented disease progression per radiological evidence or death from any cause
Overall Survival | 36 months
  Time from the date of first infusion until the date of death from any cause.
Duration of Response | 36 months
  Time from the date of the first response complete response (CRC) or partial response (PR) to the earliest date of disease progression or death from any cause. DOR is only defined for subjects who have best overall response of CR or PR

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Agensys, Inc.
Locations (21):
- United States (18):
  - Site US00012, Los Angeles, California
  - Site US00019, Stanford, California
  - Site US00017, Aurora, Colorado
  - Site US00006, New Haven, Connecticut
  - Site US00007, Miami, Florida
  - Site US00008, Tampa, Florida
  - Site US00004, Fairway, Kansas
  - Site US00005, Ann Arbor, Michigan
  - Site US00003, Detroit, Michigan
  - Site US00021, Las Vegas, Nevada
  - Site US00018, New York, New York
  - Site US00002, New York, New York
  - Site US00023, Chapel Hill, North Carolina
  - Site US00013, Philadelphia, Pennsylvania
  - Site US00020, Pittsburgh, Pennsylvania
  - Site US00024, Fairfax, Virginia
  - Site US00009, Madison, Wisconsin
  - Site US00015, Milwaukee, Wisconsin
- Canada (3):
  - Site CA00011, Calgary, Alberta
  - Site CA00001, Edmonton, Alberta
  - Site CA00010, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/ASG-22CE-13-2/
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14534&tenant=MT_AST_9011